CLINICAL TRIAL: NCT05209685
Title: Effect of Blood Flow Restriction Resistance Exercise on Functional Mobility in Pre-Frail Older Adults
Brief Title: Blood Flow Restriction on Functional Mobility in Pre-frail Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng Kung University (Other)
Responsible Party: Principal Investigator, Pei-Yun Lee, Associate professor, National Cheng Kung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A-BR-110-075
Record Dates: First submitted 2022-01-10; First posted 2022-01-26 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Frailty
Keywords: pre-frail, blood flow restriction, functional mobility
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Resistance exercise with blood flow restriction
  Interventions: Other: Resistance exercise on the lower extremities with blood flow restriction
- Control (Active Comparator): Traditional resistance exercise
  Interventions: Other: Resistance exercise on the lower extremities

INTERVENTIONS:
Other: Resistance exercise on the lower extremities — Resistance exercise mainly on the lower extremities will be executed by carrying weight according to each participant's tolerance while performing certain movements, such as side step-up, sit-to-stand, and tip-toe-standing.
  Arms: Control
Other: Resistance exercise on the lower extremities with blood flow restriction — Blood flow restriction on the thigh of the dominant leg will be used in combination with resistance exercise.
  Arms: Experimental

SUMMARY:
This study investigates the effect of blood flow restriction with resistance exercise on functional mobility in pre-frail older adults. It is hypothesized that receiving resistance exercise with blood flow restriction will exhibit better improvement on functional mobility than only receiving resistance exercise in pre-frail older adults.

DETAILED DESCRIPTION:
Participants aged over 65 years old with less than two items positive of Fried frailty phenotype assessment result will be recruited. The participants will be randomly assigned to two training groups, blood flow restriction resistance exercise and traditional resistance exercise. Both groups will receive the training 30 minutes/session, two sessions/week for six weeks. Muscle strength of the lower extremities and functional mobility tests will be used to assess outcomes at pre-training, 3-week after training, post-training, and one-month and two-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 65 years old
* Fried frailty index fulfill 1-2 criteria
* Able to walk 6 meters independently
* Able to understand and follow ≥ 3 instructions

Exclusion Criteria:

* Severe hypertension (>180/110mmHg)
* Peripheral neuropathy
* History of deep-vein thrombosis (DVT)
* Cardiovascular diseases (i.e. Heart failure NYHA Classification III or IV, myocardial infarction, pulmonary hypertension, coronary artery stenosis)
* Neuromuscular diseases (i.e. Stroke, Parkinsons' disease)
* History of resisted exercise training program within the last 6 months before screening

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 54 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change of Timed-Up and Go (TUG) test | Before intervention, 3 and 6 weeks after intervention, and one- and two-month follow ups after intervention
  Timed-Up and Go test
Change of 30 seconds sit to stand | Before intervention, 3 and 6 weeks after intervention, and one- and two-month follow ups after intervention
  30 seconds sit to stand test
Change of muscle strength of the lower extremities | Before intervention, 3 and 6 weeks after intervention, and one- and two-month follow ups after intervention
  Muscle strength of bilateral hip flexors, knee extensors, ankle dorsiflexors and plantarflexors

SECONDARY OUTCOMES:
Change of one-repetition maximum | Before intervention, 3 and 6 weeks after intervention, and one- and two-month follow ups after intervention
  One-repetiton maximum of side step-ups
Change of muscle mass | Before intervention, 3 and 6 weeks after intervention, and one- and two-month follow ups after intervention
  Muscle mass of the upper and lower extremities and trunk
Change of hand grip strength | Before intervention, 3 and 6 weeks after intervention, and one- and two-month follow ups after intervention
  Bilateral grip strength

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physical Therapy, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No